CLINICAL TRIAL: NCT07217834
Title: Effects of a Glycerol-Electrolyte Beverage on Fluid Balance in Healthy Euhydrated Men and Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: PEP-2511
Record Dates: First submitted 2025-10-08; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Fluid Balance
Keywords: hydration; electrolytes; glycerol; beverage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Beverage (Placebo Comparator): Base beverage, no electrolytes, no glycerol
  Interventions: Other: Placebo beverage, kiwi-strawberry flavor
- Experimental Beverage (Experimental): Glycerol beverage with electrolytes
  Interventions: Other: Experimental glycerol beverage, kiwi-strawberry flavor

INTERVENTIONS:
Other: Placebo beverage, kiwi-strawberry flavor — 3 equal aliquots totaling 1 liter over a 30 min period, finishing each aliquot within 5 min followed.
  Arms: Placebo Beverage
Other: Experimental glycerol beverage, kiwi-strawberry flavor — 3 equal aliquots totaling 1 liter over a 30 min period, finishing each aliquot within 5 min followed.
  Arms: Experimental Beverage

SUMMARY:
Glycerol and sodium are osmotically-active ingredients that promote fluid retention via renal water reabsorption. The purpose of this study is to compare the effects of a glycerol-electrolyte beverage on fluid balance in healthy euhydrated men and women

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* If female, subject is not pregnant
* Subject is 18-50 years of age, inclusive
* Subject is at least recreationally active (engaged in light to moderate intensity, intermittent, or steady-state exercise at least 3 days per week for at least 30 min at a time)
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study (e.g., diuretics, laxatives, weight loss drugs)
* Subject has no health conditions that would interfere with the study (e.g. cardiovascular, renal, or metabolic diseases)
* Subject is not allergic to fuji apple pear flavoring
* Subject is not allergic to Stevia
* Subject is willing to avoid alcohol consumption 24 hours prior to visits
* Subject is willing to fast overnight (~8-10 hours) prior to visits
* Subject is willing to refrain from vigorous exercise for 24 hours
* Subject is willing to eat the exact same food the day prior to each study session.
* Willing and able to provide signed informed consent to participate in the study and to comply with all study procedures and scheduled visits.

Exclusion Criteria:

* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 3 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Fluid balance | Through study completion, average of 3 weeks
  Calculated as change in nude body mass, %

SECONDARY OUTCOMES:
Fluid Balance | Through study completion, average of 3 weeks
  Calculated as change in nude body mass, kg
Urine Mass | Through study completion, average of 3 weeks
  (g)
Beverage Hydration Index | Through study completion, average of 3 weeks
  calculated as the cumulative urine mass after drinking the placebo divided by the cumulative urine mass after drinking the test beverage
Urine specific gravity | Through study completion, average of 3 weeks
  (au)
Blood Pressure | Through study completion, average of 3 weeks
  systolic/diastolic (mmHg)
Heart Rate | Through study completion, average of 3 weeks
  bpm
Subjective measures of thirst, gastrointestinal discomfort, lightheadedness and headache | Through study completion, average of 3 weeks
  Rated on a 100-pt scale from none to extreme/severe for headache, lightheaded, stomach upset, nausea, abdominal discomfort, stomach fullness, thirsty, and hydrated.
Menstrual categorization | Reported by female subjects one time at screening visit.
  Menstrual categorization chart (Elliott-Sale, 2023). Current status (e.g., contraception, regular periods or not, etc.).
Adverse Events | Through study completion, average of 3 weeks.
  Documented changes in health and symptoms. Documented both in clinic and between visits in a provided paper log reviewed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, Principal Investigator — PepsiCo R&D/Gatorade and Sports Science Institute
Locations (1):
- IMG Academy/GSSI Bradenton Gatorade Sports Science Institute, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No